CLINICAL TRIAL: NCT01082692
Title: A Phase I, Open Label Study to Evaluate the Safety, Tolerability and Immunogenicity of PENNVAX™-B (Gag, Pol, Env) + Electroporation in HIV-1 Infected Adult Participants
Brief Title: Study of PENNVAX™-B (Gag, Pol, Env) + Electroporation in HIV-1 Infected Adult Participants
Acronym: HIV-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIV-001
Record Dates: First submitted 2010-03-05; First posted 2010-03-08 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: HIV-1 Infection; HIV Infections
Keywords: HIV Infection; DNA vaccine; Electroporation; HIV therapeutic vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 3mg DNA/dose (Experimental): Subjects will receive a 4 dose series of PENNVAX-B containing 3mg of DNA/dose administered via IM injection + electroporation at Day 0, Week 4, Week 8 and Week 16.
  Interventions: Biological: PENNVAX-B

INTERVENTIONS:
Biological: PENNVAX-B — DNA plasmids delivered via IM injection + electroporation using CELLECTRA device

SUMMARY:
DNA vaccines consist of small pieces of DNA also known as plasmids, and have several potential advantages over traditional vaccines. Thus far, DNA vaccines appear to be well tolerated in humans. We have developed DNA vaccine, PENNVAX-B, which includes plasmids targeting the gag, pol, and env proteins of HIV-1. The vaccine will be delivered via electroporation (EP) which uses the CELLECTRA constant current device to deliver a small electric charge following injection, since animal studies have shown that this delivery method increases the immune response to vaccine. The vaccine will be given to HIV-1 infected subjects whose viral load is undetectable on a HAART regimen, with CD4 lymphocyte count above 400 cells/µL of blood. It is hypothesized that PENNVAX-B + EP will be safe and well tolerated.

DETAILED DESCRIPTION:
A single group of approximately 12 HIV-infected subjects will receive a 4 dose series of PENNVAX-B containing 3 mg of DNA/dose at study entry (Day 0), Week 4, 8, 16 and will be followed for a total of 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* On a stable HAART regimen for ≥3 months before the time of enrollment
* CD4-+ lymphocyte count ≥400 cells/μL on two occasions within 60 days of enrollment
* HIV-1 < 75 copies/mL on two occasions within 60 days of enrollment
* Body mass index (BMI) ≤30 kg/m^2
* Laboratory values obtained within 30 days prior to study entry:

  * Hemoglobin > 9 g/dL (female subjects) > 9.5 g/dL (male subjects)
  * Absolute neutrophil count > 1000 cells/μL
  * Platelet count > 75,000/μL
  * ALT, AST and alkaline phosphatase < 2.5 x upper limit of normal range
  * Total bilirubin < 2.5 x upper limit of the laboratory normal range
  * Serum creatinine <1.5 mg/dL X upper limit of normal (ULN)
* Female subjects of reproductive potential must have a negative serum pregnancy test performed within 30 days of initiating the protocol-specified vaccination and a negative urine pregnancy test at Day 0 (enrollment)
* Ability and willingness of subject or legal guardian/representative to give written informed consent

Exclusion Criteria:

* Any active or past AIDS-defining illness with the exception of minimal (less than 10 lesions) cutaneous Kaposi's sarcoma
* History of a CD4+ T-cell count ≤200/μL
* Grade 2 or higher CPK laboratory result
* Use of any known immunomodulatory therapy within 4 weeks prior to study entry
* Any malignancy requiring systemic or local toxic chemotherapy. Local radiation will be allowed
* Pregnancy or breast-feeding
* Uncontrolled diabetes mellitus
* Major organ transplantation
* Active alcohol or substance abuse or psychiatric illness, which in the opinion of the investigator will interfere with adherence to study requirements
* Clinically significant neurological disorder occurring within 1 year prior to study entry
* Use of systemic corticosteroids for 4 weeks within 3 months prior to study entry
* Presence of any chronic disease that in the opinion of the investigator might affect subject safety
* History of previous vaccination with an HIV-1 vaccine except where documentation of placebo is available
* History of cardiac arrhythmia
* History or evidence of autoimmune disease
* Allergies to bupivacaine or similar anesthetic
* Metal implants at the site of injection
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (i.e. infections disease) illness
* Any other conditions judged by the investigator that would limit the evaluation of a subject

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | Day 0 through Week 48
  Frequency and severity of local and systemic reactogenicity signs and symptoms, laboratory measures of safety, including CD4 and HIV RNA viral load changes, and adverse and serious adverse events.

SECONDARY OUTCOMES:
T-cell responses | Day 0 through Week 48
  Magnitude of HIV-specific immune response as determined by ELISpot assay measured two weeks following the 4th vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Tebas, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States